CLINICAL TRIAL: NCT07080710
Title: A Clinical Study on Immediate Implant Placement in the Premaxilla With Flapless Guided Surgery, Hard and Soft Tissue Augmentation and Immediate Provisionalization
Brief Title: State of the Art Immediate Implant Placement in the Premaxilla
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Ghent (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ONZ-2025-0174
Record Dates: First submitted 2025-06-23; First posted 2025-07-23 (Actual); Last update posted 2025-11-18 (Actual); Status verified 2025-11

CONDITIONS: Bone Resorption
Keywords: dental implant, single-tooth; Immediate; connective tissue graft; socket grafting; intact alveolus; non-intact alveolus
MeSH Terms: conditions — Bone Resorption

STUDY DESIGN:
Intervention Model Description: Prospective cohort study
Masking Description: As this prospective study concerns a surgical intervention, patients and treating clinicians can not be masked.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Immediate implant placement (Experimental): State of the art immediate implant placement with socket grafting and soft tissue augmentation.
  Interventions: Procedure: Immediate implant placement

INTERVENTIONS:
Procedure: Immediate implant placement — Immediate implant placement with socket grafting and soft tissue augmentation. In cases with a buccal dehiscence >3mm only this technique is applied. In cases with a buccal dehiscence between 4-6mm a collagen membrane is applied prior to socket grafting. In cases with a buccal dehiscence > 6 mm, a collagen membrane is also applied and a mixture of C-DBBM and autogenous bone chips (1:1 ratio) is used as grafting material.

SUMMARY:
The goal of this clinical study is to learn how well immediate implant placement works in the front upper jaw (premaxilla) when using flapless guided surgery, hard and soft tissue augmentation, and immediate provisional crowns. It will also learn about the safety and esthetic results of this treatment approach.

The main questions it aims to answer are:

Primary:

How much buccal bone thickness remains one year after implant placement 1mm below the implant shoulder?

Secondary:

* How do patients rate pain, healing, and esthetics after treatment?
* Are there any complications over the course of five years?
* How much buccal bone thickness remains one year after implant placement 3mm and 5mm below the implant shoulder?
* Marginal bone loss at one-year and five-year follow-up?
* Peri-implant health at one-year and five-year follow-up?
* Soft tissue changes at one-year and five-year follow-up?

Researchers will compare treatment results in patients with intact bone sockets to those with damaged (non-intact) sockets.

Participants will:

* Receive a dental implant and temporary crown on the same day as the tooth extraction
* Undergo guided, flapless surgery with bone and soft tissue grafting
* Take antibiotics and anti-inflammatories for 4 days after surgery
* Visit the clinic at 1 week, 3 months, 1 year, and 5 years for follow-up exams
* Have X-rays, digital scans, and photos taken to measure bone and soft tissue changes
* Answer questions about pain and esthetic satisfaction

DETAILED DESCRIPTION:
Preoperative three-dimensional radiograph and intra-oral digital impression:

Required to select eligible patients. All three-dimensional radiographs will be taken with lip retractors.

An intra-oral digital impression of the maxilla will also be taken. Designated software will be used to merge dicoms files (three-dimensional radiograph) and the STL file (intra-oral digital impression) to fabricate a surgical guide.

Surgery:

All surgeries will be performed by two implant surgeons . Patients start to take systemic antibiotics (Amoxicilline 1g) and anti-inflammatory medication (Ibuprofen 600 mg) 1h pre-operatively. Following local anesthesia and oral disinfection the failing tooth is extracted as atraumatically as possible and without raising a flap. Following wound debridement, a cutting implant is installed in an optimal 3D position using a surgical guide. Socket grafting is performed with collagen-enriched deproteinized bovine bone mineral to limit buccal bone resorption and to optimize soft tissue stability. Thereupon, a free gingival graft is harvested from the palatal mucosa in the premolar area and de-epithelialized to arrive at a connective tissue graft (CTG) between 1 mm and 2 mm thickness. Height and length are tailored to the dimensions of the site. Then, the CTG is sutured with two or three single sutures onto the buccal mucosa. Finally, a healing abutment is installed, which is replaced by a provisional implant crown 2 days later. Following provisional crown installation, an intra-oral radiograph is taken. This postoperative intra-oral radiograph is standard in clinical practice, also for patients who are not participating in the study.

When dealing with a shallow non-intact socket (buccal dehiscence < 3 mm = type IIa), the same technique is applied. When dealing with a dehiscence between 4 mm and 6 mm (type IIb), a collagen membrane is applied prior to socket grafting to separate the grafting material from the buccal mucosa. When dealing with a very deep dehiscence (> 6 mm = type IIc), a collagen membrane is also applied and a mixture of C-DBBM and autogenous bone chips (1:1 ratio) is used as grafting material.

Postoperative care:

Patients continue the intake of antibiotics (2 times per day) and anti-inflammatory medication (2 times per day) for 4 days and use a chlorhexidine mouth rinse during 1 week. Sutures are removed 1 week after surgery. At that time point the patient will be asked how many analgesics had been taken, and also the pain intensity will be rated on a numeric rating scale.

These are study-specific evaluations.

Three months after implant installation an intra-oral radiograph is taken to assess osseointegration. This intra-oral radiograph is standard in clinical practice, also for patients who are not participating in the study.

When the implant is successfully integrated, the patient is sent to the general dentist for fabrication of the permanent crown.

1-year registrations:

* Patients' esthetic satisfaction will be assessed on the basis of a numeric rating scale.
* A CBCT will be taken to assess buccal bone thickness at 1 mm, 3 mm and 5 mm below the implant shoulder.
* An intra-oral radiograph is taken to assess marginal bone loss.
* Peri-implant health as clinically assessed on the basis of probing depth, bleeding on probing and plaque.
* Clinical pictures to assess the esthetic outcome of the soft tissues surrounding the crown.
* An intra-oral digital impression will be taken of the upper jaw. The pre-op impression and the one-year impression will be superimposed in designated software to calculate soft tissue changes.

  5-year registrations:
* Patients' esthetic satisfaction will be assessed on the basis of a numeric rating scale.
* An intra-oral radiograph is taken to assess marginal bone loss.
* Peri-implant health as clinically assessed on the basis of probing depth, bleeding on probing and plaque.
* Clinical pictures are taken to assess the esthetic outcome of the soft tissues surrounding the crown.
* An intra-oral digital impression will be taken of the upper jaw. The pre-op impression and the five-year impression will be superimposed in designated software to calculate soft tissue changes.

ELIGIBILITY:
Inclusion Criteria:

* At least 20 years old
* Good oral hygiene defined as full-mouth plaque score ≤ 25%
* Presence of one or more incisors, cuspids or premolars in the maxilla that need to be extracted for any reason with at least one neighboring tooth present
* At least 3 mm bone available at the apical or palatal aspect of the alveoli as assessed on a three-dimensional radiograph to ensure primary implant stability
* Written informed consent.

Exclusion Criteria:

* Pregnancy (will be explicitly asked)
* Systemic diseases
* Smoking; suppuration
* > 1 mm gingival asymmetry between the failing teeth and contralateral teeth
* Failing teeth outside the bone envelop as assessed on a three-dimensional radiograph
* Untreated periodontal disease; untreated caries lesions.

Min Age: 20 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2025-07-01 (Actual); Primary Completion 2027-02-01 (Estimated); Study Completion 2032-02-01 (Estimated)

PRIMARY OUTCOMES:
Buccal bone thickness -1 (mm) | moment of enrollment and 1-year
  Buccal bone thickness at 1 mm below the implant shoulder at one-year follow-up as assessed on a three-dimensional radiograph.

SECONDARY OUTCOMES:
Patient reported outcomes | one week after surgery
  One week after surgery, patients will be asked how many analgesics have been taken. In addition, they will be asked to rate postoperative pain on a numeric rating scale (0-10).
Pink Esthetic Score | enrollment, 1-year, 5-year
  Pink Esthetic Score (PES) is registered by a trained and blinded examiner using frontal and occlusal clinical pictures taken at 1 year and 5-year follow-up. The PES results in a score from 0 (worst esthetic outcome) to 14 (perfect esthetic outcome).
Buccal bone thickness -3 and -5 (mm) | enrollment and 1-year
  Buccal bone thickness at 3mm and 5mm below the implant shoulder at one-year follow-up as assessed on a three-dimensional radiograph.
Marginal bone loss | 1-, 5-year
  Changes in the distance from the implant-abutment interface to the first bone-to-implant contact (so-called marginal bone level) at the mesial and distal aspect of each implant as measured on 2D intra-oral radiographs.
Peri-implant health | 1-, 5-year
  Peri-implant health is clinically assessed on the basis of probing depth, bleeding on probing and plaque.
Soft tissue changes | enrollment, 1-year , 5-year
  An intra-oral digital impression will be taken of the upper jaw. The pre-op impression and the one-year impression will be superimposed in designated software to calculate soft tissue changes.

CONTACTS AND LOCATIONS:
Locations (2):
- Belgium (2):
  - Ghent University, Ghent, East Flanders
  - Bv Dr. Cosyn, Zottegem, East Flanders

IPD SHARING:
Plan to Share IPD: Undecided
If the data can be included in a meta-analysis upon request by the authors, they can be transferred

REFERENCES:
- [Background] Pitman J, Christiaens V, Callens J, Glibert M, Seyssens L, Blanco J, Cosyn J. Immediate implant placement with flap or flapless surgery: A systematic review and meta-analysis. J Clin Periodontol. 2023 Jun;50(6):755-764. doi: 10.1111/jcpe.13795. Epub 2023 Mar 5. PMID 36843361
- [Background] Ickroth A, Christiaens V, Pitman J, Cosyn J. A Systematic Review on Immediate Implant Placement in Intact Versus Non-Intact Alveolar Sockets. J Clin Med. 2025 Apr 3;14(7):2462. doi: 10.3390/jcm14072462. PMID 40217911
- [Background] Furhauser R, Florescu D, Benesch T, Haas R, Mailath G, Watzek G. Evaluation of soft tissue around single-tooth implant crowns: the pink esthetic score. Clin Oral Implants Res. 2005 Dec;16(6):639-44. doi: 10.1111/j.1600-0501.2005.01193.x. PMID 16307569
- [Background] Botticelli D, Berglundh T, Lindhe J. Hard-tissue alterations following immediate implant placement in extraction sites. J Clin Periodontol. 2004 Oct;31(10):820-8. doi: 10.1111/j.1600-051X.2004.00565.x. PMID 15367183
- [Background] Assaf JH, Assaf DD, Antoniazzi RP, Osorio LB, Franca FM. Correction of Buccal Dehiscence During Immediate Implant Placement Using the Flapless Technique: A Tomographic Evaluation. J Periodontol. 2017 Feb;88(2):173-180. doi: 10.1902/jop.2016.160276. Epub 2016 Sep 13. PMID 27620655
- [Background] Barone A, Toti P, Marconcini S, Derchi G, Saverio M, Covani U. Esthetic Outcome of Implants Placed in Fresh Extraction Sockets by Clinicians with or without Experience: A Medium-Term Retrospective Evaluation. Int J Oral Maxillofac Implants. 2016 Nov/Dec;31(6):1397-1406. doi: 10.11607/jomi.4646. PMID 27861667